CLINICAL TRIAL: NCT05768880
Title: Phase 1 Study of B7-H3, EGFR806, HER2, And IL13-Zetakine (Quad) CAR T Cell Locoregional Immunotherapy For Pediatric Diffuse Intrinsic Pontine Glioma, Diffuse Midline Glioma, And Recurrent Or Refractory Central Nervous System Tumors
Brief Title: Study of B7-H3, EGFR806, HER2, And IL13-Zetakine (Quad) CAR T Cell Locoregional Immunotherapy For Pediatric Diffuse Intrinsic Pontine Glioma, Diffuse Midline Glioma, And Recurrent Or Refractory Central Nervous System Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BrainChild-04
Record Dates: First submitted 2023-02-17; First posted 2023-03-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma; Recurrent CNS Tumor, Adult; Recurrent, CNS Tumor, Childhood; Refractory Primary Malignant Central Nervous System Neoplasm
Keywords: CNS Tumor; DIPG; DMG; B7-H3; HER2; IL13-zetakine; EGFR806; CAR T cell; pediatric; brain tumor
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma; Central Nervous System Neoplasms; Recurrence; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - DIPG (Experimental)
  Interventions: Biological: SC-CAR4BRAIN
- Arm B - DMG & recurrent/refractory tumors (Experimental)
  Interventions: Biological: SC-CAR4BRAIN

INTERVENTIONS:
Biological: SC-CAR4BRAIN — Courses of weekly intraventricular CNS administered SC-CAR4BRAIN infusions for 3 weeks, then 1 week off

SUMMARY:
This is a Phase 1 study of central nervous system (CNS) locoregional adoptive therapy with SC-CAR4BRAIN, an autologous CD4+ and CD8+ T cells lentivirally transduced to express to express combinations of B7-H3, EGFR806, HER2, and IL13-zetakine chimeric antigen receptors (CAR). CAR T cells are delivered via an indwelling catheter into the ventricular system in children and young adults with diffuse intrinsic pontine glioma (DIPG), diffuse midline glioma (DMG), and recurrent or refractory CNS tumors.

A child or young adult meeting all eligibility criteria, including having a CNS catheter placed into their ventricular system, and meeting none of the exclusion criteria will have their T cells collected. The T cells will then be bioengineered into a second-generation CAR T cell that target B7H3, EGFR806, HER2, and IL13-zetakine on tumor cells.

Patients will be assigned to 1 of 2 treatment Arms based on the type of their tumor:

* Arm A is for patients with DIPG (meaning primary disease localized to the pons, metastatic disease is allowed) anytime after standard radiation OR after progression.
* Arm B is for patients with non-pontine DMG (meaning DMG in other parts of the brain such as the thalamus or spine) anytime after standard radiation OR after progression. This Arm also includes other recurrent/refractory CNS tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must be age ≥ 1 and ≤ 26 years (except for the first 3 subjects, who must be age ≥ 12 and ≤ 26 years).
2. Subject disease classified as one of the following:

   1. DIPG at any timepoint following completion of standard radiotherapy
   2. DMG at any timepoint following completion of standard radiotherapy
   3. Evidence of refractory or recurrent CNS disease for which there is no routine therapy, defined by either of the following:

   i. New site or sites of measurable or evaluable disease by radiographic imaging or histologic confirmation following completion of routine care first-line therapy for which curative salvage therapy is not available or amenable, OR ii. Measurable or evaluable disease that persists following completion of routine care first-line therapy for which curative salvage therapy is not available or amenable
3. Able to tolerate apheresis or already has an apheresis product available for use in manufacturing
4. CNS reservoir catheter, such as an Ommaya or Rickham catheter, present in the proper location for CNS-directed therapy delivered as specified for BrainChild-04
5. Life expectancy ≥ 8 weeks
6. Lansky or Karnofsky score ≥ 60.
7. If patient does not have previously obtained apheresis product, patient must have discontinued, and recovered from acute toxic effects of, all prior chemotherapy, immunotherapy, and radiotherapy and discontinue the following prior to enrollment:

   * ≥ 7 days post last chemotherapy/biologic therapy administration
   * 3 half lives or 30 days, whichever is shorter post last dose of anti-tumor antibody therapy
   * Must be at least 30 days from most recent cellular infusion
   * All systemically administered corticosteroid treatment therapy must be stable or decreasing within 1 week prior to enrollment with maximum dexamethasone dose of 2.5 mg/m2/day. Corticosteroid physiologic replacement therapy is allowed.
8. Adequate organ function
9. Adequate laboratory values
10. Subjects of childbearing/fathering potential must agree to use highly effective contraception from the time of enrollment through 12 months following the last T cell infusion

Exclusion Criteria:

1. Presence of ≥ Grade 3 cardiac dysfunction or symptomatic arrhythmia requiring intervention
2. Presence of primary immunodeficiency/bone marrow failure syndrome
3. Presence of clinical and/or radiographic evidence of impending herniation in the CNS
4. For Arm A subjects only: Presence of > Grade 3 dysphagia
5. Presence of active malignancy other than the CNS tumor under study
6. Presence of active severe infection, defined as either of the following:

   1. Positive blood culture within 48 hours of enrollment, OR
   2. Fever > 38.2ºC AND clinical signs of infection within 48 hours of enrollment
7. Pregnant or breastfeeding
8. Subject and/or authorized legal representative unwilling to provide consent/assent for study participation, including participation in the 15-year follow-up period, which is required if CAR T cell therapy is administered
9. Presence of any condition that, in the opinion of the investigator, would prohibit the subject from undergoing treatment under this protocol

Ages: 1 Year to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2028-01-15 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
Manufacturing Feasibility | 42 days
  Number and percent of subjects with sufficient therapeutic product generated to receive two courses on the intended dose regimen
Safety of SC-CAR4BRAIN | 28 days post-final SC-CAR4BRAIN infusion
  Establish the safety, defined by the adverse events of fractionated intraventricular CNS administration of adoptive therapy with SC-CAR4BRAIN in children and young adults with DIPG, DMG, or recurrent/refractory CNS tumors
Dose level | 28 days
  Establish the maximally tolerated dose regimen (MTDR) and recommended Phase 2 dose regimen (RP2DR) of fractionated intraventricular CNS administered SC CAR4BRAIN infusions.
Administration feasibility | 98 days
  Number of subjects meeting criteria for their initial CAR T infusion and number of subjects meeting criteria for at least 2 courses of CAR T infusions

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Ronsley, MD, Study Chair — Seattle Children's Hospital; Rebecca Ronsley, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No